CLINICAL TRIAL: NCT04971265
Title: Cognitive Interviewing of Survey Items for a Computer Adaptive Test of Parent Knowledge and Beliefs
Brief Title: Family Supports and Beliefs Survey
Acronym: FSBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB21-0355
Record Dates: First submitted 2021-06-28; First posted 2021-07-21 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Beliefs About Child Development

STUDY DESIGN:
Intervention Model Description: Participants are randomized to see one of four scenarios at the start of the study, while taking the Family Supports and Beliefs Survey [#1: LowSES, High Societal Supports; #2, Low SES, Low Societal Supports; #3 High SES, High Societal Supports; or #4 High SES, Low Societal Supports]
Who Masked: Participant
Masking Description: Participants will not know that there are 3 other scenarios within the Family Supports and Beliefs survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low SES/High Supports (Experimental): Participants assigned to the "Low SES/High Supports" arm will see the "Low SES/High Supports" intervention
  Interventions: Behavioral: Low SES/High Supports
- Low SES/Low Supports (Experimental): Participants assigned to the "Low SES/Low Supports" arm will see the "Low SES/Low Supports" intervention
  Interventions: Behavioral: Low SES/ Low Supports
- High SES/High Supports (Experimental): Participants assigned to the "High SES/High Supports" arm will see the "High SES/High Supports" intervention
  Interventions: Behavioral: High SES/High Supports
- High SES/Low Supports (Experimental): Participants assigned to the "Low SES/High Supports" arm will see the "High SES/Low Supports" intervention
  Interventions: Behavioral: High SES/Low Supports

INTERVENTIONS:
Behavioral: Low SES/High Supports — Participant will read the following scenario: Michael and Kim are a young couple living with their 2-year-old child. Michael works as a janitor in a residential building, while Kim works as a cashier in a supermarket. Where they live, all parents have 12 weeks of paid parental leave, access to free full-day center-based daycare for children aged 0 to 3, free full-day preschool for children aged 3 to 5 (early education programs to prepare for kindergarten), and free parenting classes.
  Arms: Low SES/High Supports
Behavioral: Low SES/ Low Supports — Participants will read the following scenario: Michael and Kim are a young couple living with their 2-year-old child. Michael works as a janitor in a residential building, while Kim works as a cashier in a supermarket. Where they live, parents have 1 week of paid parental leave, full-day center-based daycare for children aged 0 to 3 is available for around $900 per month, full-day preschool for children aged 3 to 5 (early education programs to prepare for kindergarten) is available for around $1400 a month, and they can take parenting classes for $50 per hour.
  Arms: Low SES/Low Supports
Behavioral: High SES/High Supports — Participants will read the following scenario: Michael and Kim are a young couple living with their 2-year-old child. Michael works as a lawyer in a private company, while Kim works as a manager at a bank. Where they live, all parents have 12 weeks of paid parental leave, access to free full-day center-based daycare for children aged 0 to 3, free full-day preschool for children aged 3 to 5 (early education programs to prepare for kindergarten), and free parenting classes.
  Arms: High SES/High Supports
Behavioral: High SES/Low Supports — Participants will read the following scenario: Michael and Kim are a young couple living with their 2-year-old child. Michael works as a lawyer in a private company, while Kim works as a manager at a bank. Where they live, parents have 1 week of paid parental leave, full-day center-based daycare for children aged 0 to 3 is available for around $900 per month, full-day preschool for children aged 3 to 5 (early education programs to prepare for kindergarten) is available for around $1400 a month, and they can take parenting classes for $50 per hour.
  Arms: High SES/Low Supports

SUMMARY:
Participants will complete a survey (The Family Supports and Beliefs Survey), which will measure their existing beliefs about the role of societal resources in supporting families and young children. Participants will randomly see one of four fictional scenarios and then be asked questions related to that scenario as well as items related to stress and self-efficacy. We hypothesize that the type of scenario a participant is presented with before taking a survey may affect how they answer subsequent questions.

This survey is being administered as part of a broader project designed to test items that are being developed for a new measure, the Survey of Parent/Provider Expectations and Knowledge Computer Adaptive Test (SPEAK CAT).

ELIGIBILITY:
Inclusion Criteria:

* Must live in the United States

Exclusion Criteria:

* Individuals who cannot complete the survey in English
* Individuals under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Beliefs about the role of parenting and family supports on child development | At enrollment only
  As measured by the Family Supports and Beliefs Survey

SECONDARY OUTCOMES:
Stress and self-efficacy | At enrollment only
  As measured by the Family Supports and Beliefs Survey

CONTACTS AND LOCATIONS:
Overall Officials: Dana Suskind, M.D., Principal Investigator — University of Chicago
Locations (1):
- TMW Center for Early Learning + Public Health at the University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the Family Supports and Beliefs survey will be made available upon request for replication purposes.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified data will be made available upon request, after publication of the results
Access Criteria: Access will be granted for replication purposes

DOCUMENTS (1):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT04971265/Prot_001.pdf